CLINICAL TRIAL: NCT05725369
Title: The Effects of Combined Lifestyle Intervention (CLI) in Patients With Inflammatory Bowel Disease (IBD)
Acronym: GLI-IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-16137
Record Dates: First submitted 2023-01-10; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: lifestyle; diet; combined lifestyle intervention; exercise
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Combined Lifestyle Intervention (CLI) — In the Netherlands, the combined lifestyle intervention (CLI, in Dutch: gecombineerde leefstijlinterventie (GLI)) is available for all Dutch citizens with a BMI ≥ 30 mg/kg2 or a BMI between 25 and 30 mg/kg2 and an increased risk of diabetes or cardiovascular disease. The CLI aims to realize health benefits for people with a moderate weight-related health risk and consists of a two-year program with advice and counseling to improve health-related behavior such as physical activity and diet.

SUMMARY:
A single-center observational study to investigate the effects of combined lifestyle intervention (CLI, in Dutch: gecombineerde leefstijlinterventie, GLI) in patients with Inflammatory Bowel Disease.

DETAILED DESCRIPTION:
This is an exploratory observational study of IBD patients ≥ 18 years old with a BMI ≥ 30 mg/kg2 or a BMI between 25 and 30 and an increased risk of diabetes or cardiovascular disease, who are or have been referred to the CLI.

During the 2-year CLI program, fitness measurements take place according to CLI protocol and by the CLI provider: bodyweight, BMI, waist circumference, fat percentage and the EQ-5D-5L are recorded at baseline and 1-year and 2-year timepoints. Whilst patients are offered a CLI referral, willingness to partake will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Diagnosis of IBD (Ulcerative Colitis, Crohn's Disease or IBD-Unclassified) confirmed by clinical, endoscopic, and histological evidence prior to screening as per standard criteria;
* BMI ≥ 30 mg/kg2 or a BMI between 25 and 30 mg/kg2 and an increased risk of diabetes or cardiovascular disease;
* Patients that are or have been referred to the CLI;
* Oral informed consent must be obtained and documented in EPIC.

Exclusion Criteria:

* Serious underlying disease other than IBD that in the opinion of the investigator may interfere with the subject's ability to participate fully in the study or would compromise subject safety (such as major neurological disorders, certain orthopedic impairments or any unstable, uncontrolled or severe systemic medical disorder);
* If female, the subject is pregnant or lactating;
* Illiteracy (disability to read and understand Dutch).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old with a BMI ≥ 30 mg/kg2 or a BMI between 25 and 30 mg/kg2 and an increased risk of diabetes or cardiovascular disease, who are eligible to be referred to the CLI or have already been referred to the CLI.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in bodyweight | 2 years
  Measured in kilograms
Decrease in BMI | 2 years
  Measures in mg/kg2
Decrease in waist circumference | 2 years
  Measured in centimeters
Decrease in fat percentage | 2 years
  Measured in percentages
Quality of life | 2 years
  EQ-5D-5L score

SECONDARY OUTCOMES:
Adherence | 2 years
  Adherence to the CLI (i.e. amount of patients to stop the CLI prematurely)
Willingness | 2 years
  Willingness to partake in the CLI (and to be referred to the CLI)
IBD related adverse events | 2 yera
  Incidence of IBD related adverse events during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Marjolijn Duijvestein, MD PhD, Principal Investigator — Radboud University Medical Center (Radboudumc)

IPD SHARING:
Plan to Share IPD: Undecided